CLINICAL TRIAL: NCT06484140
Title: Evaluation of the Financial Navigation Program for Improving Financial Toxicity Among Breast Cancer in China
Brief Title: Financial Navigation Program for Improving Financial Toxicity Among Breast Cancer in China
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xiaoyi Yuan, Principal Investigator, Fudan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: XYuan2312288-16
Record Dates: First submitted 2024-06-26; First posted 2024-07-03 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2024-06

CONDITIONS: Breast Neoplasm Female; Financial Toxicity; Financial Navigation
MeSH Terms: conditions — Financial Stress

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Financial Navigation (Experimental): Participants will receive financial navigation service, including
  * Needs Assessment: provide a brief introduction of cancer-related FT and assess patients' information needs using a self-made cost-related health literacy questionnaire;
  * Cost-Related Health Education: mainly include topics regarding communication of cost, treatment-related cost, health insurance policies, and family support;
  * Resource and Service Referral: promote timely referral to financial assistance programs and clinical professionals when identify unaddressed problems;
  * Personalized Counseling Module: provide one-on-one counseling for symptom management, cost-related issues, and coping strategies.
  Interventions: Behavioral: Financial Navigation
- Usual Care (Active Comparator): Participants will receive usual care during hospitalization and regular follow-up after discharge. Participants have the freedom to utilize any financial resources, but financial navigators do not offer comprehensive information support. When participants actively inquire about cancer treatment-related costs or financial planning strategies, financial navigators will answer their questions.
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: Financial Navigation — During hospitalization, participants will receive needs assessment, and one-on-one cost-related health education with a material booklet. Resource and service referral will be delivered face-to-face or by phone when the navigator identifies unaddressed problems. Within three months after discharge, participants will receive monthly follow-up phone calls and personalized counseling via WeChat.
  Arms: Financial Navigation
Other: Usual Care — Participants will receive usual oncology care during hospitalization and regular follow-up after discharge. Participants have the freedom to utilize any financial resources, but financial navigators do not offer comprehensive information support.
  Arms: Usual Care

SUMMARY:
The goal of this study is to access the impact of a financial navigation program on improving financial toxicity among patients with breast cancer in China.

The main questions it aims to answer are:

* Does the intervention alleviate participants' financial toxicity?
* Does the intervention enhance participants' cost-related health literacy?
* Does the intervention improve participants' shared decision-making?
* Does the intervention reduce participants' perceived stress?

Researchers will compare the financial navigation program with usual oncology care to evaluate its effectiveness.

Participants will receive the comprehensive financial navigation, including:

* Needs assessment;
* Cost-related health education, mainly including topics regarding communication of cost, treatment-related cost, health insurance policies, and family support;
* Resource and service referral;
* Personalized counseling.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed with breast cancer and undergoing surgery during this admission;
* Female, age 18 years or older;
* Receiving or expected to receive one or more of the following therapies: chemotherapy, radiotherapy, endocrine therapy, targeted therapy, and immunotherapy;
* Eastern Cooperative Oncology Group Performance Status 0-2;
* Provided informed consent to participate in this study.

Exclusion Criteria:

* Diagnosed with ductal carcinoma in situ (DCIS)
* Presence of any serious psychiatric disorders;
* Cognitive impairments;
* Difficulty in reading, writing, or communicating in Chinese.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2024-06-17 (Actual); Primary Completion 2024-11-11 (Actual); Study Completion 2024-11-17 (Actual)

PRIMARY OUTCOMES:
Financial toxicity | Baseline, 1st month and 3rd month since baseline
  Financial toxicity will be measured with the Comprehensive Score for Financial Toxicity-Functional Assessment of Chronic Illness Therapy Version 2 (COST-FACIT-V2); lower scores (range, 0-44) indicating greater financial toxicity.
Material domain of financial toxicity | 1st month and 3rd month since baseline
  Material domain of financial toxicity will be measured with 2 items adapted from the Medical Expenditure Panel Survey (MEPS).
Behavioral domain of financial toxicity | 1st month and 3rd month since baseline
  Behavioral domain of financial toxicity will be measured by employment changes and cost-related nonadherence with 6 items adapted from MEPS and previous literature.

SECONDARY OUTCOMES:
Cost-related health literacy | Baseline, 1st month and 3rd month since baseline
  The cost-related health literacy will be measured with homemade 10-item questionnaire, with higher scores indicating higher cost-related health literacy.
Shared decision-making | Baseline, 1st month and 3rd month since baseline
  The shared decision-making ability will be measured with 9-item shared decision-making questionnaire (SDM-Q-9); higher scores (range, 0-45) indicating a greater degree of participants' involvement in shared decision-making.
Perceived stress | Baseline, 1st month and 3rd month since baseline
  The perceived stress will be measured with Perceived Stress Scale (PSS); higher scores (range, 0-56) indicating greater perceived stress.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
We do not plan to share individual participant data due to privacy concerns and confidentiality agreements with participants.